CLINICAL TRIAL: NCT05071937
Title: Phase ll Study of a BET Inhibitor, ZEN003694, Combined With a PARP Inhibitor, Talazoparib, in Patients With Recurrent Ovarian Cancer
Brief Title: ZEN003694 Combined With Talazoparib in Patients With Recurrent Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alexander B Olawaiye, MD (Other)
Collaborators: Pfizer (Industry); Zenith Epigenetics (Industry)
Responsible Party: Sponsor-Investigator, Alexander B Olawaiye, MD, Professor, Department of Obstetrics, Gynecology & Reproductive Sciences, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 21-091
Record Dates: First submitted 2021-09-27; First posted 2021-10-08 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: PARP enzyme; bromodomain and extra terminal domain (BET) proteins
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZEN003694 + Talazoparib (Experimental): ZEN003694: 48.0 mg daily (oral) in 28-day cycles
  Talazoparib: 0.75 mg daily (oral) at the same time as ZEN003694
  Interventions: Drug: ZEN003694; Drug: Talazoparib

INTERVENTIONS:
Drug: ZEN003694 — ZEN003694 has shown promising activity in the treatment of solid tumors and hematologic (blood) cancers by reducing the multiplication of cancer cells.
Drug: Talazoparib — Talazoparib kills cancer cells by inhibiting and trapping the enzyme PARP, which is known to be involved in the development of many types of cancers.

SUMMARY:
This Phase 2, open label, study with safety lead in of oral talazoparib in combination with ZEN003694 given daily in 28-day cycles will enroll patients with recurrent ovarian, fallopian tube or primary peritoneal carcinoma.

DETAILED DESCRIPTION:
This study aims to determine how effective the combination of ZEN003694 and talazoparib is based on how patients respond. ZEN003694 (and developed by Zenith Epigenetics Ltd.) has shown promising activity in the treatment of solid tumors and hematologic (blood) cancers by reducing the multiplication of cancer cells. Talazoparib is an extremely effective drug being developed for the treatment of a variety of human cancers. Talazoparib kills cancer cells by inhibiting and trapping the enzyme PARP, which is known to be involved in the development of many types of cancers. These two drugs are not FDA approved in the treatment of ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Females age ≥ 18 years (at time of signing informed consent)
2. ECOG status 0 or 1
3. Pathologically documented ovarian, fallopian tube, or primary peritoneal carcinoma.
4. Prior therapy with PARPi either as maintenance or therapeutic settings.
5. All recurrent ovarian cancer both platinum sensitive and platinum resistant are allowed.
6. Any prior number of cancer therapy regimens
7. Measurable disease per RECIST 1.1
8. Known BRCA1/2 status
9. Adequate laboratory parameters at Screening including:

   1. Hemoglobin ≥ 9.0 gm/dL without transfusions during the 4 weeks prior to Screening
   2. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
   3. Platelet count ≥ 150,000/mm3
   4. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.0 x ULN or if liver function abnormalities due to liver metastases AST and ALT ≤ 5.0 x ULN
   5. Total bilirubin ≤ 1.5 x ULN (≤ 3.0 x ULN for subjects with known Gilbert's syndrome)
   6. Serum Creatinine ≤ 1.5 X ULN
   7. Prothrombin time (PT), international normalized ratio (INR) and partial thromboplastin time (PTT) < 1.5 x ULN
10. Female subjects may be enrolled if they are not of childbearing potential, permanently sterile or who are post-menopausal, defined as no menses for at least 1 year without an alternative medical cause and FSH levels in the post-menopausal range. Female subjects of childbearing potential may be enrolled if they consistently and correctly use a highly effective form of contraception. Highly effective forms of contraception include: combined (estrogen and progestogen hormonal contraceptives (oral, intravaginal, transdermal) associated with inhibition of ovulation; progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomized partner; sexual abstinence. Female subjects should not donate eggs from the time point of study drug administration until at least 7 months thereafter
11. Females of childbearing potential must have a negative serum pregnancy test before the first dose of study drug and must agree to serum pregnancy tests during the study.
12. Females may not be breast-feeding at the first dose of study drug, during study participation or through 7 months after the last dose of study drug.
13. Ability to swallow capsules and comply with study procedures.
14. Ability to understand and willingness to sign informed consent form prior to initiation of any study procedures.
15. Patients with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to study enrollment, have discontinued corticosteroid treatment for these metastases for at least 4 weeks and are neurologically stable with evidence of no disease progression for 6 months.

    Exclusion Criteria:
16. Current or anticipated use of medications known to be strong inhibitors or inducers of CYP3A4 or substrates of CYP1A2 with narrow therapeutic windows. Strong inhibitors, inducers or substrates must be discontinued at least 7 days prior to the first administration of study drug.
17. Current or anticipated use within 7 days prior to the first administration of study drug, or during the study, of strong P-gp inhibitors.
18. Use of oral Factor Xa inhibitors (i.e., rivaroxaban, apixaban, betrixaban, edoxaban otamixaban, letaxaban, eribaxaban) and Factor IIa inhibitors (i.e., dabigatran). Low molecular weight heparin is allowed
19. Radiation to >25% of the bone marrow
20. Treatment with a bone-targeted radionuclide within 6 weeks of first dose of study drug
21. Prior chemotherapy or radiation within 3 weeks of study enrollment
22. Have previously received an investigational BET inhibitor (including previous participation in studies with Zenith drug, ZEN003694)
23. QTcF interval > 470 msec
24. Insufficient recovery from prior treatment-related toxicities except for alopecia, fatigue and Grade 2 neuropathy
25. Non-healing wound, ulcer or bone fracture (not including a pathological bone fracture caused by a pre-existing pathological bone lesion)
26. Brain metastases not adequately treated and/or clinically stable (at the discretion of the Investigator) for at least 6 months prior to the start of study treatment.
27. Patients with ovarian carcinosarcoma
28. Known impaired cardiac function or clinically significant cardiac disease such as uncontrolled supraventricular arrhythmia, ventricular arrhythmia requiring therapy, or congestive heart failure (New York Heart Association functional class III or IV)
29. Myocardial infarction or unstable angina within 6 months prior to the first administration of study drug
30. Known myelodysplastic syndrome
31. Other clinically significant co-morbidities, such as uncontrolled pulmonary disease, active central nervous system disease, active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy, or any other condition that could compromise safety or the patient's participation in the study
32. Impairment of gastrointestinal function that may significantly alter the absorption of ZEN003694 or talazoparib
33. Other known active cancer requiring therapy at time of study entry or that progressed or required treatment within 3 years prior to starting study drug (except for skin basal cell carcinoma or squamous cell carcinoma or in situ cervical cancer)
34. History of infection with (screening tests not required): human immunodeficiency virus; hepatitis B virus with currently active disease defined as hepatitis B surface antigen (HBsAg) positivity; or hepatitis C virus unless previously treated and viral load is undetectable except following situations:

    * HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of enrollment are eligible for this trial.
    * Patients with a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection are allowed to be included if: participant on a stable dose of antiviral therapy, HBV viral load below the limit of quantification. HCV viral load below the limit of quantification.
35. Major surgery other than diagnostic surgery, dental surgery or stenting within 4 weeks prior to the first administration of study drug
36. Concurrent participation in another clinical investigational treatment trial
37. Any other reason that in the opinion of the Investigator would prevent the patient from completing participation or following the study schedule

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2033-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response | Up to 48 months
  Confirmed complete response or partial response by RECIST 1.1. Per RECIST v1.1. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Adverse events at least possibly related to treatment | Up to 48 months
  Adverse Events which occur from first day of treatment, characterized by type, grade and relatedness to treatment according to CTCAE v5.0, considered to be possibly, probably or definitely related to study treatment.
Duration of Response | Up to 48 months
  Time from start of response to documented disease progression by RECIST v1.1 or death due to any cause. Progression as defined by RECIST v1.1 for target lesions: Progressive Disease (PD): smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). For non-target lesions:
  Progressive Disease (PD): Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Progression-free survival (PFS) | Up to 6 years
  Time from first response to to treatment until documented disease progression by RECIST v1.1 or death due to any cause. Progression as defined by RECIST v1.1 for target lesions: Progressive Disease (PD): smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). For non-target lesions:
  Progressive Disease (PD): Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Overall survival (OS) | Up to 6 years
  Overall survival (OS), defined as time from first dose of study treatment until death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander B Olawaiye, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No